CLINICAL TRIAL: NCT03750357
Title: Percutaneous Electrical Nerve Stimulation (PENS) of the Auricle for Acute Pain Management Post Cardiac Surgery
Brief Title: Percutaneous Electrical Nerve Stimulation (PENS) of the Auricle for Post Operative Pain Solution(POPS) - Cardiac Surgery
Acronym: POPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DyAnsys, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PR2-POPS-18; CS/PRv2.0/01/2018 (Other: Dyansys India)
Record Dates: First submitted 2018-11-17; First posted 2018-11-23 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2018-11

CONDITIONS: Post Operative Pain; Midline Sternotomy Incision
Keywords: Cardiac surgery pain reduction; Post operative pain; PENS; Neurostimulation
MeSH Terms: conditions — Pain, Postoperative | interventions — Implantable Neurostimulators

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Relief v 2.0 with Paracetamol (Experimental): Group A will be treated with Primary Relief v 2.0(1 - 100Hz) sweep stimulation with increase in power of the stimulation for fixed interval of time.
  Interventions: Device: Primary Relief v 2.0
- Only Paracetamol (No Intervention): Group B will be treated with paracetamol drug.

INTERVENTIONS:
Device: Primary Relief v 2.0 — To prove the effectiveness of Post Operative Pain Solution using Primary relief v 2.0 by Percutaneous Electrical Nerve Stimulation in the auricle.
  Other Names: Neurostimulator
  Arms: Primary Relief v 2.0 with Paracetamol

SUMMARY:
Percutaneous Electrical Nerve Stimulation (PENS) of the auricle for acute pain management post cardiac surgery

DETAILED DESCRIPTION:
A well formulated analgesic protocol is fundamental to fast tracking post cardiac surgery. Traditional analgesic methods have their own set of drawbacks unique to cardiac surgery. Opioids have well established side effects like nausea, vomiting, respiratory depression, urinary retention. Regional anesthetic techniques in anti coagulated patients may result in potentially catastrophic neurological, bleeding and thromboembolic sequelae. Non steroidal Anti Inflammatory Drugs (NSAIDs) have been associated with increased cerebrovascular events, renal dysfunction, sternal wound infections. These make alternative therapies, including non pharmacological modalities, attractive options for optimal analgesic therapy during the post operative period.

Alternative methods like topical application of COX -2 inhibitors, intravenous magnesium, Transcutaneous Electrical Nerve Stimulation (TENS) have been tried with varied results in cardiac surgery. A somatotopic relationship has been described between the auricle and the other anatomical regions of the body. When specific points are accurately identified along the meridians of the ear and stimulated electrically, analgesic effects are known to occur. Percutaneous Electrical Nerve Stimulation (PENS) of the auricle and its efficacy in management of post midline sternotomy pain has not been evaluated previously. Primary Relief v 2.0 is a device which provides continuous PENS aimed at non pharmacological post operative pain management.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery patient with midline sternotomy incision

Exclusion Criteria:

1. Thoracotomy incisions
2. Patients with pacemakers,
3. Post operative cognitive dysfunction
4. Anticipated ventilation > 24 hrs
5. Pre operative opioid therapy
6. Ear infections
7. Skin lesions / allergy to adhesive materials
8. Re-exploration for any reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2018-11-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
PAIN Relief by physical examination by HCP | After 2 hours of device activation
  Relief of pain when the dosage of the anesthesia level gradually decreases after the surgery completion. This is measured by physical interaction with the patient by the health care provider.

CONTACTS AND LOCATIONS:
Overall Officials: Rohini M Balaji, MBBS., DNB, Principal Investigator — Sri Jayadeva Institue of Cardiovascular Science and Research
Locations (1):
- Sri Jayadeva Institute of cardiovascular Science and Research, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No